CLINICAL TRIAL: NCT04287595
Title: Inhalation Aromatherapy on Nausea, Vomiting and Anxiety During Autologous Hematopoietic Stem Cell Transplantation: An Open-label Randmized Controlled Trial
Brief Title: Effect of Orange Aroma on Nausea, Vomiting and Anxiety During Autologous Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nur Izgu, Assoc. Prof., RN, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Nausea; Vomiting; Anxiety State
Keywords: anxiety; hematopoietic stem cell transplantation; inhalation aromatherapy; nausea; randomized controlled trial
MeSH Terms: conditions — Nausea; Vomiting; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): inhalation aromatherapy with orange essential oil
  Interventions: Other: Inhalation aromatherapy with orange essential oil
- control group (No Intervention): routine care

INTERVENTIONS:
Other: Inhalation aromatherapy with orange essential oil
  Arms: intervention group

SUMMARY:
Patients undergoing stem cell transplantation for the first time will be entered. Participants will be randomized to one of two study arms: Arm 1: intervention (routine care+ inhalation aromatherapy); Arm 2: Control (Routine care) Hypotheses: (1) Patients receiving inhalation aromatherapy will experience less severe nausea and less frequent vomiting episodes than those receiving only routine care; and (2) patients receiving inhalation aromatherapy will demonstrate lower anxiety levels just after AHSCT than those receiving only routine care.

DETAILED DESCRIPTION:
Earlier research indicates that aromatherapy is promising to relieve in DMSO related nausea and anxiety in autologous stem cell transplant patients. The current study seeks to confirm and extend these findings in a 2-arm, open-label randomized, controlled study of 70 cancer patients undergoing autologous stem cell transplantation. All patients will receive a standardized premedication. Arm 1: Intervention (inhalation aromatherapy with orange essential oil during stem cell infusion); Arm 2: Control (routine care). The researchers hypothesize that inhalation aromatherapy with orange essential oil will be effective in reducing DMSO related nausea and vomiting and demonstrate lower anxiety levels just after autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* the absence of any mental conditions including depression, anxiety disorders, psychotic disorders or dementia that may affect the patients' communication abilities

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease or asthma,
* a history of allergy to orange or orange essential oil,
* presence of persistent nausea and vomiting due to conditioning regimens,
* receiving antiemetic other than routine premedication,
* patients undergoing AHSCT for the second or more time were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-28 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Change in nausea severity | At 1st minute of each stem cell infusion bag
  Patient report Nausea severity will be assessed based on patient report by using a visual analog scale. The patients will be asked to rate their nausea severity and place a mark on the scale from 0 to 10.
change in number of vomiting | From 1st minute of the stem cell infusion to completion of the intervention
  Observation Number of vomiting and retching episodes will be observed by the researcher who apply aromatherapy and recorded in a vomiting and retching episodes form.

SECONDARY OUTCOMES:
anxiety | Through stem cell infusion completion, an avarege of 30 minutes
  Patient report State Anxiety Inventory will be used to measure anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Izgu, PhD, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No